CLINICAL TRIAL: NCT02191254
Title: A 12-week, Double-blind, Randomised, Placebo-controlled, Multicentre Trial to Evaluate Efficacy and Tolerability of Antistax® Film Coated Tablets, 360 mg/Day Orally, in Male and Female Patients Suffering From Chronic Venous Insufficiency
Brief Title: Efficacy and Tolerability of Antistax® in Male and Female Patients Suffering From Chronic Venous Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1138.4
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Antistax

ARMS (2):
- Antistax® (Experimental): 1 tablet per day for 12 weeks
  Interventions: Drug: Antistax®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Antistax®
  Arms: Antistax®
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the efficacy and tolerability of Antistax® film-coated tablets in patients with chronic venous insufficiency (CVI, Clinical condition, Etiology, Anatomic location, Pathophysiology (CEAP) Classification: Clinical Class 3, or 4a)

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* CVI, Clinical Class 3 (oedema) or 4a (mild skin changes ascribed to venous disease, e.g. pigmentation), according to the CEAP classification
* Willing and able to give written informed consent prior to participation in the study

Exclusion Criteria:

Concomitant diseases:

* Decompensated cardiac insufficiency
* Oedema not due to venous disease of the legs (e.g., latent cardiac insufficiency, renal insufficiency, lymphoedema, etc)
* Peripheral arterial disease (ankle/arm pressure index < 0.9)
* Current acute phlebitis or thrombosis
* Renal insufficiency (serum creatinine > 1.5 mg/dl)
* Liver disease (SGPT > 3x upper limit of normal)
* Other diseases: hyper- or hypocalcaemia, malignancies
* Anamnestic indications of diabetic microangiopathy or polyneuropathy
* Drug and/or alcohol abuse
* Severe climacteric complaints: changes in, or initiation with post-menopausal hormone replacement therapy within the last 3 months
* Immobility
* Avalvulia
* Klippel-Trénaunay-Weber-Syndrome (Naevus varicosis osteohypertrophicus, Haemangiectasia hypertrophicans)
* State after pulmonary embolism
* Recognised hypersensitivity to the trial drug ingredients
* Current florid venous ulcus
* Clinical indication for a necessary, specific phlebologic acute treatment, e.g. compression treatment, phlebectomy, etc.

Previous treatments:

* Patients who are on compression therapy and/or are wearing support stockings and who optimally benefit from these measures
* Treatment with venous drugs within the last 2 weeks prior to the intake of study medication
* Changes in or unstable response to treatment with theophylline, diuretics, cardiac glycosides, ACE inhibitors, calcium antagonists, or laxatives within the last 2 weeks prior to the intake of study medication

Concomitant treatment/non-drug therapy exclusion criteria:

* Other venous drugs apart from the trial medication
* Venous surgery or sclerotherapy within the last 12 month at the leg used for volumetry
* Extensive use of laxatives
* Major surgery requiring full anaesthesia

Other exclusion criteria:

* Previously studied under this protocol
* Participation in another clinical trial within the previous 90 days or during the present study
* Patient is investigator, co-investigator, or study nurse in this study
* Pregnant or nursing women or inadequate birth control methods (this applies to females of childbearing potential only)
* Patients considered as mentally ill as well as unable to work or with limited working ability, or unable (or only partially able) to follow the spoken or written explanations concerning the trial
* Patients in a bad general health state according to the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2004-04; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in limb volume determination | Baseline, day 84
  water displacement method

SECONDARY OUTCOMES:
Changes in limb volume determination | Baseline, day 21 and day 42
  water displacement method
Changes in the calf circumference | Baseline, at day 21, 42 and 84
  in centimeters
Changes in the ankle circumference | Baseline, at day 21, 42, and 84
  in centimeters
Changes in the subjective symptoms of CVI measured by Visual Analogue Scales (VAS) | Baseline, at day 21, 42, and 84
Global assessment of efficacy by the patient on a 4-point verbal rating scale (VRS) | day 84
Global assessment of efficacy by the investigator on a 4-point VRS | day 84
Global assessment of tolerability by the patient on a 4-point VRS | day 84
Global assessment of tolerability by the investigator on a 4-point VRS | Day 84
Number of patients with adverse events | up to 12 weeks
Number of patients with clinically significant changes in laboratory values | Baseline, week 12
Number of patients with clinically significant changes in vital signs (Blood Pressure (BP), Pulse Rate (PR)) | Baseline, up to 12 weeks

REFERENCES:
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449